CLINICAL TRIAL: NCT03150719
Title: Phase 3b, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Safety, Efficacy, and Tolerability of Tezacaftor/Ivacaftor (TEZ/IVA) in an Orkambi-experienced Population Who Are Homozygous for the F508del CFTR Mutation
Brief Title: A Study to Evaluate Safety, Efficacy, and Tolerability of TEZ/IVA in Orkambi® (Lumacaftor/Ivacaftor) -Experienced Subjects With Cystic Fibrosis (CF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX16-661-114; 2017-000540-18 (EudraCT Number)
Expanded Access: NCT03278314 (Approved for marketing)
Record Dates: First submitted 2017-05-03; First posted 2017-05-12 (Actual); Results first posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — tezacaftor, ivacaftor drug combination; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo matched to TEZ/IVA fixed-dose combination tablet orally once daily in the morning followed by placebo matched to IVA tablet orally once daily in the evening for 56 days.
  Interventions: Drug: Placebo
- TEZ/IVA (Experimental): Participants received TEZ 100 milligram (mg)/IVA 150 mg fixed-dose combination tablet orally once daily in the morning and IVA 150 mg tablet orally once daily in the evening for 56 days.
  Interventions: Drug: Tezacaftor/Ivacaftor; Drug: Ivacaftor

INTERVENTIONS:
Drug: Tezacaftor/Ivacaftor — TEZ 100 mg/IVA 150 mg fixed-dose combination tablet.
  Other Names: TEZ/IVA; VX-661/VX-770
  Arms: TEZ/IVA
Drug: Ivacaftor — IVA 150 mg tablet.
  Other Names: VX-770; IVA
  Arms: TEZ/IVA
Drug: Placebo — Placebo matched to TEZ/IVA fixed-dose combination tablet.
  Arms: Placebo
Drug: Placebo — Placebo matched to IVA tablet.
  Arms: Placebo

SUMMARY:
Study VX16-661-114 (Study 114) is a Phase 3b, randomized, double-blind, placebo-controlled, parallel-group, multicenter study in subjects aged 12 years and older with CF who are homozygous for the F508del mutation on the cystic fibrosis transmembrane conductance regulator gene (CFTR) gene and who discontinued treatment with Orkambi due to respiratory symptoms considered related to treatment. This study is designed to evaluate the safety and efficacy of Tezacaftor/Ivacaftor (TEZ/IVA).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with scheduled visits, treatment plan, study restrictions, laboratory tests, contraceptive guidelines, and other study procedures.
* Prior discontinuation of Orkambi, with at least 1 respiratory sign or symptom considered related to therapy.
* Resolution or stabilization of qualifying event(s) >28 days prior to Screening.
* Discontinuation of Orkambi therapy must have occurred within approximately 12 weeks from the first dose of Orkambi.
* Homozygous for F508del mutation in the CFTR gene as documented in the subject's medical record. If genotype documentation is not available in the medical record, genotyping will be performed during screening.
* FEV1 ≥25% and ≤90% of predicted normal for age, sex, and height.
* Stable CF disease as judged by the investigator.
* Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

* History of any comorbidity that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject.
* Recent rapid or progressive deterioration in respiratory status.
* Receiving continuous oxygen at >2L/min or on face-mask ventilation.
* Any protocol-defined exclusionary laboratory values at Screening.
* Child-Pugh Class B or C hepatic impairment.
* An acute upper or lower respiratory infection, pulmonary exacerbation, or change in therapy for pulmonary disease within 28 days before Day 1.
* Documentation of colonization with organisms associated with a more rapid decline in pulmonary status.
* History of lung transplantation since most recent initiation of Orkambi.
* History of alcohol or drug abuse in the past year as deemed by the investigator.
* Participation in an investigational drug study or use of a CFTR modulator within 28 days or 5 terminal half-lives of the investigational drug or modulator (whichever is longer).
* Use of restricted medications or foods within the specified window before the first dose of study drug, or an anticipated need or use of restricted medication or foods after the first dose of study drug.
* Pregnant or nursing females: Females of child-bearing potential must have a negative pregnancy test at Screening and Day 1.
* Other protocol defined exclusion criteria could apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (53):
- United States (41):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - UCSF - Fresno, Community Regional Medical Center, Fresno, California
  - Miller Children's Hospital / Long Beach Memorial, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Rady Children's Hospital, San Diego, California
  - National Jewish Health, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Central Florida Pulmonary Group, Orlando, Florida
  - Arnold Palmer Hospital, Orlando, Florida
  - Tampa General Hospital Cardiac and Lung Transplant Clinic, Tampa, Florida
  - Children's Speciality Services at North Druid Hills, Atlanta, Georgia
  - St. Luke's CF Center of Idaho, Boise, Idaho
  - Advocate Children's Hospital - Park Ridge / North Suburban Pulmonary and Critical Care Consultants, Niles, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - The University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kentucky Clinic, Lexington, Kentucky
  - Tulane Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital Cystic Fibrosis Center, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Billings Clinic, Billings, Montana
  - Mount Sinai Beth Israel, New York, New York
  - New York Medical College, Valhalla, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Santiago Reyes, M.D., Oklahoma City, Oklahoma
  - Drexel University College of Medicine/ Drexel Adult Cystic Fibrosis Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Tennessee Medical Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah / Primary Children's Medical Center, Salt Lake City, Utah
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Children's Hospital of Richmond at VCU, Children's Pavilion, Richmond, Virginia
- France (7):
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Hospitalier Universitaire De Grenoble - Hopital Michallon, Grenoble
  - CHU de Montpellier - Hopital Arnaud de Villeneuve, Montpellier
  - Centre Hospitalier Universitaire De Nantes, Nantes
  - Centre hospitalier universitaire de Nice, Pulmonology, Nice
  - Hopital Cochin, Paris
  - Centre Hospitalier Universitaire - Hopitaux de Rouen, Rouen
- Germany (5):
  - Charite Paediatric Pulmonology Department, Berlin
  - Ruhrlandklinik Westdeutsches Lungenzentrum am Klinikum Essen, Essen
  - Klinikum Innenstadt, University of Munich, München
  - Pneumologische Praxis Pasing, München
  - Universitaetsklinikum Tuebingen Klinik fuer Kinder- und Jugendmedizin, Tübingen

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 98 participants were randomized: 47 in placebo group and 51 in tezacaftor (TEZ)/ivacaftor (IVA) group. One participant in TEZ/IVA group did not receive any study drug.
Period: Overall Study
Arm/Group | Placebo | TEZ/IVA
Started | 47 | 50
Completed | 46 | 48
Not Completed | 1 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Death | 0 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- TEZ/IVA: Participants received TEZ 100 mg/IVA 150 mg fixed-dose combination tablet orally once daily in the morning and IVA 150 mg tablet orally once daily in the evening for 56 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | TEZ/IVA | Total
Number analyzed (Participants) | 47 | 50 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (10.0) | 34.3 (8.7) | 33.8 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 31 | 61
  Male | 17 | 19 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 40 | 41 | 81
  Unknown or Not Reported | 4 | 8 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 42 | 42 | 84
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Respiratory Adverse Events of Special Interest (RAESIs)
Description: RAESIs included chest discomfort, dyspnea (shortness of breath), respiration abnormal (chest tightness), asthma, bronchial hyperreactivity, bronchospasm, and wheezing.
Time Frame: Day 1 up to Day 84
Population: Safety set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEZ/IVA
Number analyzed (Participants) | 47 | 50
Participants | 10 | 7

2. Secondary Outcome: Absolute Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) at Average of Day 28 and Day 56 Measurements
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: Baseline, Day 28 and Day 56
Population: Full analysis set (FAS) included all randomized participants who carried the intended cystic fibrosis transmembrane conductance regulator gene (CFTR) allele mutation and had received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: percent predicted of FEV1
Arm/Group | Placebo | TEZ/IVA
Number analyzed (Participants) | 47 | 50
percent predicted of FEV1 | -0.6 (3.4) | 2.2 (4.8)
Statistical Analysis 1: Comparison: Placebo vs TEZ/IVA; Test type: Superiority; Mean Difference = 2.7, 95% CI 2-sided [1.0 to 4.4]

3. Secondary Outcome: Relative Change From Baseline in ppFEV1 at Average of Day 28 and Day 56 Measurements
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: Baseline, Day 28 and Day 56
Population: FAS.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | TEZ/IVA
Number analyzed (Participants) | 47 | 50
percent change | -1.5 (8.1) | 5.2 (12.0)
Statistical Analysis 1: Comparison: Placebo vs TEZ/IVA; Test type: Superiority; Mean Difference = 6.7, 95% CI 2-sided [2.5 to 10.9]

4. Secondary Outcome: Absolute Change From Baseline in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score at Average of Day 28 and Day 56 Measurements
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: Baseline, Day 28 and Day 56
Population: FAS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TEZ/IVA
Number analyzed (Participants) | 47 | 50
units on a scale | 4.7 (15.4) | 5.7 (14.2)
Statistical Analysis 1: Comparison: Placebo vs TEZ/IVA; Test type: Superiority; Mean Difference = 1.1, 95% CI 2-sided [-4.9 to 7.0]

5. Secondary Outcome: Tolerability as Assessed by Number of Participants Who Discontinued Treatment
Time Frame: Day 1 through Day 56
Population: Safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEZ/IVA
Number analyzed (Participants) | 47 | 50
Participants | 2 | 2

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Day 84
Population: Safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEZ/IVA
Number analyzed (Participants) | 47 | 50
Participants
  Participants with AEs | 39 | 37
  Participants with SAEs | 9 | 5

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 84
Arm/Group | Placebo | TEZ/IVA
All-Cause Mortality (participants affected / at risk) | 0/47 | 1/50
Serious Adverse Events (participants affected / at risk) | 9/47 | 5/50
Other Adverse Events (participants affected / at risk) | 28/47 | 30/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=47) | TEZ/IVA (N=50)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 7 | 3
Sepsis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=47) | TEZ/IVA (N=50)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Abdominal pain upper (Gastrointestinal disorders) | 5 | 4
Constipation (Gastrointestinal disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Nasopharyngitis (Infections and infestations) | 0 | 6
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 9 | 4
Headache (Nervous system disorders) | 7 | 6
Bacterial test positive (Investigations) | 0 | 3
Fatigue (General disorders) | 4 | 2
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT03150719/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/19/NCT03150719/SAP_001.pdf